CLINICAL TRIAL: NCT01776736
Title: Study of Posture Correction Girdle of Adolescents With Early Scoliosis
Brief Title: Safety and Efficacy of Posture Correction Girdle for Adolescent With Early Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Joanne Yip, Lecturer, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITF-237-11
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Posture correction
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Posture Correction Girdle (Experimental): Posture Correction Girdle applied for 8 hours per day. Clinical, radiographic, and self-report follow-up within the girdling period (6 months).
  Interventions: Device: Posture Correction Girdle

INTERVENTIONS:
Device: Posture Correction Girdle — Posture Correction Girdle applied for 8 hours per day. Clinical, radiographic, and self-report follow-up within the girdling period (6 months).

SUMMARY:
For AIS, the caring of patients with spinal deformities has a long and varied history. Severe spinal deformities can greatly reduce pulmonary and cardiac functions, which may lead to death from cardiopulmonary failure. Therefore, surgery is generally suggested when the curvature of the spine is greater than 45-50 degrees. The adverse psychological impact of orthoses treatment on patients and its poor compliance has been a well-recognised problem. Some orthotic research studies indicate that early intervention of spinal deformities is particularly desirable. Taking into consideration current clinical practices, if the curve is less than 20 degrees, even if the child is at a high risk of progressive spinal deformity during the age of 10-16 at puberty, treatment is nothing more than just observation.

This project aims to combine clinical experience with textile and materials sciences to research and develop a posture correction girdle for adolescents with early scoliosis. As a result, this will reduce the future likelihood of brace wear or surgery.

In this study, the eligible subjects will be given tailor-made posture correction girdles to wear it 8 hours daily. Monitoring and observation will be provided during the six months girdling period. Data will be collected before and after the girdling by X-ray radiograph for analysis, in order to comparison the spine curvature condition. Locomotion of the subject with and without wearing the posture correction girdle will also be reference.

DETAILED DESCRIPTION:
For AIS, the caring of patients with spinal deformities has a long and varied history. Severe spinal deformities can greatly reduce pulmonary and cardiac functions, which may lead to death from cardiopulmonary failure. Therefore, surgery is generally suggested when the curvature of the spine is greater than 45-50 degrees. The adverse psychological impact of orthoses treatment on patients and its poor compliance has been a well-recognised problem. Some orthotic research studies indicate that early intervention of spinal deformities is particularly desirable. Taking into consideration current clinical practices, if the curve is less than 20 degrees, even if the child is at a high risk of progressive spinal deformity during the age of 10-16 at puberty, treatment is nothing more than just observation.

This project aims to combine clinical experience with textile and materials sciences to research and develop a posture correction girdle for adolescents with early scoliosis. As a result, this will reduce the future likelihood of brace wear or surgery.

The eligible subjects will be given tailor-made posture correction girdles. Monitoring and observation will be provided during the girdling period. Data will be collected before and after the girdling by X-ray radiograph for analysis, in order to comparison the spine curvature condition. Locomotion of the subject with and without wearing the posture correction girdle will also be reference.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 13 years
* Diagnosis of AIS in early stage
* Primary Cobb angle equals to or less than 20 degrees
* Pre-menarchal or post-menarchal by no more than 1 year
* Ability to read and understand English or Chinese
* At high risk for curve progression
* Skeletally immature (Risser grade 0, 1, or 2)
* Physical and mental ability to adhere to posture correction girdle protocol

Exclusion Criteria:

* Contraindications for x-ray exposure
* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
* History of previous surgical or orthotic treatment for AIS
* Contraindications for pulmonary and / or exercise tests
* Psychiatric disorders
* Recent trauma
* Recent traumatic (emotional) event

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression of the spinal curve | From baseline to 6 months
  No progression of the spinal curve (no increase of Cobb angle) by radiographic measures.

SECONDARY OUTCOMES:
Progression of the spinal curve | From baseline to 6 months
  The progression of the spinal curve within control (increase of Cobb angle < 5 degrees)
Posture improvement | From baseline to 6 months
  Improvement of posture by clinical photographs assessment

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Yip, PhD, Principal Investigator — The Hong Kong Polytechnic University; Kit-Lun Yick, Ph.D, Study Chair — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China